CLINICAL TRIAL: NCT06616272
Title: Cervical Spine Focused Treatment for Patients With Persistent Concussion Symptoms and Neck Pain: Pilot Study
Brief Title: Cervical Spine Focused Treatment for Patients With Persistent Concussion Symptoms and Neck Pain
Acronym: ConCerv
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Michael Schneider, DC, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY24040157
Record Dates: First submitted 2024-09-16; First posted 2024-09-27 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Brain Concussion; Neck Pain
Keywords: concussion care; cervical rehabilitation; neck pain
MeSH Terms: conditions — Brain Concussion; Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cervical spine focused treatment and standard concussion care (Active Comparator): The cervical spine focused treatment will start concurrently with the standard care once the participant is randomized to this group. The participants will receive early cervical spine focused treatment 2x/week for 4 weeks. In addition to the cervical spine focused treatment, this group will also receive standard concussion care interventions individualized to the participant's needs 1x/week concurrently during the same 4-week period of time. After 4 weeks, the participant will discontinue the cervical spine focused treatment but may continue with standard concussion care for an additional 4 weeks (maximum total treatment duration is 8 weeks).
  Interventions: Other: Cervical rehabilitation; Other: Standard Concussion Care
- Standard concussion care alone followed by delayed cervical spine focused treatment (Active Comparator): Participants randomized to the delayed cervical spine focused treatment group will only receive the standard concussion care (individualized to their needs) 1x/week for the initial 4 weeks. At the 4-week timepoint, the cervical spine focused treatment will be added to the standard concussion care at a frequency of twice a week for 4 weeks. Should a participant be cleared for return to activity prior to the end of the 4-week period, cervical spine focused treatment will be suspended. The maximum total treatment duration is 8 weeks; 1x/week for weeks 1-8 for the standard concussion care and 2x/week for weeks 4-8 for the cervical spine focused treatment.
  Interventions: Other: Cervical rehabilitation; Other: Standard Concussion Care

INTERVENTIONS:
Other: Cervical rehabilitation — * Manual joint mobilization (Grades I-V) of painful and restricted cervical spine segments.
  * Supine manual cervical traction to stretch and mobilize the cervical spinal tissues.
  * Manual soft tissue mobilization of the cervical, upper thoracic and/or shoulder muscles.
  * Passive stretching of hypertonic muscles and active strengthening of hypotonic muscles.
  * Motor-control and isometric exercises to activate the deep neck flexors.
Other: Standard Concussion Care — Standard Concussion Care interventions are individualized to each patient and their adjudicated profile(s)/moderating factor(s) and may include any/all of the following:
  * Behavioral regulation
  * Vestibular rehabilitation
  * Oculomotor rehabilitation
  * Exertion rehabilitation
  * Pharmacological management
  * Behavioral sleep intervention
  * *Cervical spine rehabilitation (the variable of interest in this study)
  * Psychotherapy

SUMMARY:
Assess the feasibility of recruiting, enrolling and randomizing patients with concussion symptoms and neck pain to receive manual therapy and cervical rehabilitative exercises in addition to standard concussion treatment.

In the usual care workflow provided at the participating concussion clinic, cervical spine rehab is not typically introduced until after week 4. The rationale is that neck pain is often a self-limiting condition that may resolve spontaneously, without the need for specific cervical spine rehab.

This study is chiefly focused on feasibility aims that revolve around developing changes to barriers in workflow issues at the participating concussion clinic, that would allow for earlier introduction of cervical spine rehab.

DETAILED DESCRIPTION:
This is a a single site pilot randomized controlled trial consisting of a total of 40 participants with concussion and neck pain, randomized to one of two groups (n=20 per group):

1. early cervical spine focused treatment combined with standard concussion care.
2. standard concussion care alone for 4 weeks, followed by delayed introduction (after 4 weeks) of cervical spine focused treatment (which is the usual care workflow at our clinical partner site.)

Both groups will receive the combination of cervical spine focused treatment and standard concussion care; the only variation being the timing of the introduction of the cervical spine care.

The primary endpoint will be 4 weeks from start of cervical rehabilitation intervention. The secondary would be the point of discharge. The duration of active participation in the study will be 8 weeks for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed concussion
* Patient endorses neck pain OR difficulty moving their neck (moderate or severe; score of 2 or 3 for items 16 and 25 from concussion CP screen)
* Willingness to be randomized
* 8-90 days post injury
* English Speaking

Exclusion Criteria:

* Previous concussion within the past 6 months
* Prior history of ischemic/vascular events
* Previous treatment for current symptoms
* Prior treatment for neck pain/headaches in the past year
* Workers' compensation claim and/or litigation associated with injury
* Diagnosed substance use disorder
* Prior cervical spine surgery
* Prior fracture and or dislocation/subluxation of the cervical spine
* Diagnosed inflammatory arthritis

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Enrolling 6 new participants per month
Treatment Adherence | 2 months
  Assess the rate of adherence to treatment with a goal of participant attending ≥ 75% (6 of 8) of scheduled visits.
Conversion Rate | 6 months
  Ratio of concussion patients with neck pain approached about participation or referred for screening to those actually screened. As well as conversion rate of concussion patients screened for participation to those enrolled and randomized.
Adverse Event Rate | 2 months
  Rates of expected side effects and adverse events

SECONDARY OUTCOMES:
Concussion Clinical Profile screen (CP screen) | Baseline, 4 week, 8 week
  Patient reported outcome regarding their concussion symptoms. The raw score ranges from 0 to 87. The scale helps identify specific clinical profiles and associated modifiers in concussion patients.
Numeric pain rating scale (NPRS) | Baseline, 4 week, 8 week
  Patient reported measure regarding average neck pain over past week. The score range from 0 to 10 where 0 is no pain and 10 is considered the worst pain imaginable.
Neck Disability index (NDI) | Baseline, 4 week, 8 week
  Patient reported outcome regarding their neck pain related disability. The scale ranges from 0-50 that are then converted to percentages. The scores are interpreted as: 0-20%: minimal disability; 21-40%: moderate disability; 41-60%: severe disability; and >60%: complete disability.
Pain, Enjoyment and General Activity Score (PEG) | Baseline, 4 week, 8 week
  Patient reported outcome regarding their pain and its interference to enjoyment in life and general activity in the past week. The scale has three individual items that are scored from 0 to 10. The overall score is the average of the three individual item scores rounded to the nearest whole number for clinical use.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Schneider, DC, PhD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (2):
  - UPMC sports medicine, Pittsburgh, Pennsylvania
  - Greenfield Clinic-Children's Wisconsin, Milwaukee, Wisconsin
- UPMC Sports Surgery Clinic, Dublin, Ireland
- Sports Medicine Northern Ireland, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kontos AP, Elbin RJ, Trbovich A, Womble M, Said A, Sumrok VF, French J, Kegel N, Puskar A, Sherry N, Holland C, Collins M. Concussion Clinical Profiles Screening (CP Screen) Tool: Preliminary Evidence to Inform a Multidisciplinary Approach. Neurosurgery. 2020 Aug 1;87(2):348-356. doi: 10.1093/neuros/nyz545. PMID 31950187
- [Background] Quatman-Yates CC, Hunter-Giordano A, Shimamura KK, Landel R, Alsalaheen BA, Hanke TA, McCulloch KL. Physical Therapy Evaluation and Treatment After Concussion/Mild Traumatic Brain Injury. J Orthop Sports Phys Ther. 2020 Apr;50(4):CPG1-CPG73. doi: 10.2519/jospt.2020.0301. PMID 32241234
- [Background] McCrory P, Meeuwisse WH, Aubry M, Cantu B, Dvorak J, Echemendia RJ, Engebretsen L, Johnston K, Kutcher JS, Raftery M, Sills A, Benson BW, Davis GA, Ellenbogen RG, Guskiewicz K, Herring SA, Iverson GL, Jordan BD, Kissick J, McCrea M, McIntosh AS, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator CH, Turner M. Consensus statement on concussion in sport: the 4th International Conference on Concussion in Sport held in Zurich, November 2012. Br J Sports Med. 2013 Apr;47(5):250-8. doi: 10.1136/bjsports-2013-092313. No abstract available. PMID 23479479
- [Background] McCrory PR, Ariens T, Berkovic SF. The nature and duration of acute concussive symptoms in Australian football. Clin J Sport Med. 2000 Oct;10(4):235-8. doi: 10.1097/00042752-200010000-00002. PMID 11086747
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Hurwitz EL, Carragee EJ, van der Velde G, Carroll LJ, Nordin M, Guzman J, Peloso PM, Holm LW, Cote P, Hogg-Johnson S, Cassidy JD, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Treatment of neck pain: noninvasive interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S123-52. doi: 10.1097/BRS.0b013e3181644b1d. PMID 18204386
- [Background] Reid SA, Rivett DA, Katekar MG, Callister R. Sustained natural apophyseal glides (SNAGs) are an effective treatment for cervicogenic dizziness. Man Ther. 2008 Aug;13(4):357-66. doi: 10.1016/j.math.2007.03.006. Epub 2007 Oct 22. PMID 17951095
- [Background] van der Walt K, Tyson A, Kennedy E. How often is neck and vestibulo-ocular physiotherapy treatment recommended in people with persistent post-concussion symptoms? A retrospective analysis. Musculoskelet Sci Pract. 2019 Feb;39:130-135. doi: 10.1016/j.msksp.2018.12.004. Epub 2018 Dec 11. PMID 30583251
- [Background] Jones C, Sterling M. Clinimetrics: Neck Disability Index. J Physiother. 2021 Apr;67(2):144. doi: 10.1016/j.jphys.2020.09.001. Epub 2021 Mar 19. No abstract available. PMID 33753016
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333